CLINICAL TRIAL: NCT06313983
Title: A Phase Ⅲ Randomized, Open Label, Parallel, Multicenter To Assess Efficacy and Safety Study of Hemay022 in Combination With AI In Postmenopausal HER2+/ER+ Advanced Breast Cancer Patients Treated With Trastuzumab-containing Regimens
Brief Title: A Phase Ⅲ Study of Hemay022 in Combination With AI In Advanced Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM022BC3C01; NCT05122494 (obsolete NCT alias)
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemay022 and AI (Experimental): Hemay022 in combination with AI will be taken orally once daily. Planned dose of Hemay022 will be 500mg daily for 21 days.
  Interventions: Drug: Hemay022+AI
- Lapatinib and Capecitabine (Active Comparator): lapatinib in combination with capecitabine will be taken in suitable dose until disease progression or death, etc.
  Interventions: Drug: Lapatinib+Capecitabine

INTERVENTIONS:
Drug: Hemay022+AI — hemay022：orally once daily，A 21-day cycle
  Arms: Hemay022 and AI
Drug: Lapatinib+Capecitabine — Take the pills according to the instructions
  Arms: Lapatinib and Capecitabine

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Hemay022 combined with AI (exemestane or letrozole) in the treatment of ER+/HER2+ advanced breast cancer patients based on the progression-free survival (PFS) assessed by the independent review committee (IRC). The second purpose of this study is to evaluate the pharmacokinetics and efficacy of Hemay022 in combination with AI, and the safety of Hemay022 in combination with AI.

The trial plans to recruit 339 subjects, who will be randomly divided into two cohorts (the experimental group is hemay022 combined with AI, and the control group is lapatinib combined with capecitabine). During the treatment period, imaging examinations and anti-tumor efficacy evaluations will be performed regularly until the subject develop disease progression or starts receiving other treatments or dies or refuses to come to the hospital for follow-up or the trial is terminated, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old；
2. Subjects must give informed consent to the study before the study entry and voluntarily sign a written informed consent form;
3. Breast cancer subjects diagnosed by pathology（histology or cytology）;
4. ER positive and HER2 over-expression (immunohistochemical IHC test 3+ and/or in situ hybridization ISH test positive)；Previous test results are acceptable.
5. Advanced/metastatic breast cancer that has previously received treatment failure with trastuzumab (or trastuzumab biosimilar) regimen;Or (new) adjuvant therapy during treatment with trastuzumab (or trastuzumab biosimilar) or within 12 months after the end of treatment, disease recurrence or progression；Patients with first-line systemic treatment for relapse (previously received trastuzumab or trastuzumab biosimilars)；Or patients who are not suitable for trastuzumab treatment；Patients who have failed previous anti-HER2-ADC drug therapy can also be included.
6. At least one lesion (measurable and/or non-measurable) that can be evaluated by CT/MRI and meets the reproducible evaluation requirements of RECIST V1.1;
7. ECOG Performance Status of 0-1;
8. The estimated survival time is more than 3 months;
9. Postmenopausal women

   Postmenopausal is defined as meeting any one of the following four conditions:

   Past bilateral oophorectomy; Age ≥60 years old; Age <60 years old, natural menopause ≥12 months, in the past 1 year without chemotherapy, tamoxifen, toremifene or ovarian castration, the level of follicle stimulating hormone (FSH) and estradiol Within the postmenopausal range (use the reference range of the local laboratory).

   Patients younger than 60 years old who are taking tamoxifen or toremifene, their FSH and estradiol levels are within the postmenopausal range (use the reference range of the local laboratory); Premenopausal or perimenopausal women who do not meet the above-mentioned menopausal criteria can also be included in this study, but they must also receive ovarian suppression therapy that meets the standards of medical or surgical castration treatment. Drug ovarian suppression therapy has been started at least 21 days before the start of this program, and Must be continued during the treatment plan;
10. Adequate bone marrow, liver, kidney, and coagulation Bone Marrow Function (No blood transfusion or adjuvant leukocyte or platelet augmentation drugs were used within 1 week before screening) Absolute value of neutrophils (ANC) ≥1.5×109/L Hemoglobin (HB) ≥90g/L (transfusion allowed) Platelet (PLT) ≥80×109/L Liver function Liver function grade Child-Pugh A/B (≤9 points) Alanine transferase (ALT) or aspartate aminotransferase (AST) ≤2.5 ULN in the absence of liver metastasis; ALT or AST≤ 5x ULN with liver metastasis Renal function: serum creatinine ≤1.5 times ULN;
11. All previous treatment-related toxicities must be CTCAE (version 5.0) ≤ Grade 2 at the time of randomization, except for hair loss, pigmentation, and long-term toxicity caused by radiotherapy (which cannot be recovered by the investigator's judgment)；
12. Women patients of childbearing age (including their partners) have no pregnancy plan and voluntarily take effective contraceptive measures from the signing of the informed consent form to 3 months after the last medication.

Exclusion Criteria:

1. Patients with visceral crisis（Visceral crisis is defined as the dysfunction of several organs confirmed by symptoms, signs, laboratory tests, and rapid disease progression.Visceral crisis does not simply refer to the presence of visceral metastases, but to critical visceral conditions that require rapid and effective treatment to control the disease progression, especially when the opportunity for chemotherapy is lost after progression）
2. Patients with the presence of spinal cord compression or brain, meningeal metastases
3. Patients who have been treated with a small molecule HER2 tyrosine kinase inhibitor (HER2-TKI) (medication course ≤2 weeks is excluded)
4. Have received radiotherapy within 4 weeks prior to study；
5. Have received chemotherapy for advanced breast cancer> 1 lines (the subjects who have used chemotherapy drugs must have stopped the chemotherapy drugs for ≥ 4 weeks before being enrolled in this study);
6. Patients with parenteral nutrition; malabsorption syndrome; or any condition possibly affecting drug absorption or inability to tolerate oral medications;
7. Use of any drug that inhibits or induces hepatic metabolism of Hemay022 within 2 weeks prior to study and entire study duration, for example CYP3A4 strong inhibitors or strong inducers;
8. Patients who are known to have a history of allergies to Hemay022, lapatinib、AI (letrozole, exemestane) capecitabine or similar drugs.
9. Left ventricular ejection fraction (LVEF) <50％ as measured by echocardiogram or MUGA scan.
10. Positive blood for human immunodeficiency virus (HIV antibody); Positive hepatitis B surface antigen and HBV-DNA>upper limit of normal; Active hepatitis C virus (HCV) infection
11. Patients with active infection requiring intravenous anti-infective treatment
12. Arrhythmias requiring treatment , including atrial fibrillation, supraventricular tachycardia ,ventricular tachycardia, ventricular fibrillation, or patients with coronary heart disease have symptoms requiring medicine treatment, myocardial infarction within 1 year, congestive heart failure (CHF)
13. Confirmed QTc prolongation (≥500ms) (heart rate corrected according to Bazett formula or Fridericia formula)
14. People with a history of interstitial lung disease that needs treatment, a history of radiation pneumonitis, or clinically active interstitial lung disease
15. Have received other clinical trial drugs within 4 weeks before the study
16. Major surgery or injury less than 4 weeks before the study
17. The study period must be accompanied by other antitumor therapy，such as chemotherapy, targeted therapy, hormone therapy, immunotherapy, radiotherapy (except symptomatic local radiotherapy)
18. Any other malignant cancer within 5 years with the exception of adequately treated cervical cancer in situ or basal and squamous cutaneous cell carcinomas
19. Any condition that would make the subject inappropriate for this study by the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2022-01-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival（mPFS）based on IRC assessment according to RECIST v1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS defined as the proportion of patients alive and without progression

SECONDARY OUTCOMES:
Overall Survival (OS) of the two group according to RECIST v1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  OS is defined as the time from random to any cause of death
Objective response rate ( ORR, partial response rate+ complete response rate) according to RECIST v1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  ORR defined as the proportion of subjects in complete response (CR) or (partial response) PR
Clinical benefit rate (CBR) according to RECIST v1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Clinical benefit rate defined as percentage of patients with stable disease (SD) ≥ 6 months/partial response (PR)/complete response (CR).
Duration of Response (DOR) according to RECIST v1.1 | The earliest date from the first recorded CR or PR to the first recorded disease progression or death，assessed up to 100 months
  DOR defined as the duration after the first assessment as CR or PR, only applicable to subjects who have achieved remission
Time to Response (TTR) | Start of treatment until the earliest date of CR or PR recorded for the first time，assessed up to 100 months
  TTR defined as the time from random to CR or PR for the first time

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

REFERENCES:
- [Derived] Zhang P, Wang L, Zhen Y, Wang Z, Zhang H, Jones R, Xu B. A phase I study of Hemay022, an irreversible dual EGFR/HER2 tyrosine kinase inhibitor in Chinese patients with HER2-positive advanced breast cancer. Chin J Cancer Res. 2024 Feb 29;36(1):46-54. doi: 10.21147/j.issn.1000-9604.2024.01.05. PMID 38455366